CLINICAL TRIAL: NCT01762501
Title: Azilsartan Circadian and Sleep Pressure - the 1st Study
Brief Title: Azilsartan Circadian and Sleep Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sogo Rinsho Médéfi Co., Ltd. (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACS1
Record Dates: First submitted 2012-12-18; First posted 2013-01-07 (Estimated); Results first posted 2015-12-28 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-11

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension | interventions — azilsartan; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Azilsartan (Experimental): Azilsartan 20mg/day in oral administration, single dose Treatment duration: 8 weeks
  Interventions: Drug: Azilsartan
- Amlodipine (Active Comparator): Amlodipine 5mg/day in oral administration, single dose Treatment duration: 8 weeks
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Azilsartan — Azilsartan 20mg/day
  Other Names: AZILVA Tablets
  Arms: Azilsartan
Drug: Amlodipine — Amlodipine 5mg/day
  Other Names: Amlodin Tablets etc.
  Arms: Amlodipine

SUMMARY:
To determine the efficacy of Azilsartan 20 mg versus Amlodipine 5 mg oral administration once per day for 8 weeks in patients with grade I or grade II essential hypertension.

DETAILED DESCRIPTION:
Treatment

<Run-in period> Use of any antihypertensives, including azilsartan and amlodipine, is prohibited during the run-in period.

<Treatment period> Subjects who are considered eligible for participation in the study based on the results of eligibility assessment during the run-in period will be randomized to the azilsartan 20 mg or amlodipine 5 mg group at a ratio of 1:1 according to the following stratification factors; the type of awake-sleep blood pressure variation determined based on the data from ABPM at the start of run-in, complication status (chronic kidney diseases [CKD], type 2 diabetes), age, and sex.

Subjects will start treatment with either antihypertensive after examination for the start of treatment (Week 0) and visit the study site every 2 weeks, 5 visits in total, until the end of treatment (Week 8).

Subjects will orally take azilsartan 20 mg or amlodipine 5 mg, according to their group allocation, once daily before or after breakfast in the morning.

ELIGIBILITY:
Inclusion Criteria:

* Grade I or II essential hypertension
* The sitting systolic blood pressure is in term of 140-179 mmHg, or sitting diastolic blood pressure is in term of 90-109 mmHg at the both two time points at the beginning of the observation period and at the beginning of a treatment period (Week0)
* 20 years old or older at the time of the informed consent
* Able to give written informed consent before participating in the research
* Therapeutic category during the observation period: Ambulatory

Exclusion Criteria:

* Secondary hypertension, grade III hypertension (sitting systolic blood pressure greater than or equal to 180 mmHg or sitting diastolic blood pressure greater than or equal to 110 mmHg), malignant hypertension
* More than 2 kinds of antihypertensive agents for treatment on the hypertension
* History of taking following medicines within 2 weeks before start of the observation period.

When subject with taking any of the following medicine at the time of informed consent is included, stop to take the medicine for determined period after the informed consent.

I. Antihypertensive agents II. Antianginal agents III. Antiarrhythmic agents (except single time use of the lidocaine hydrochloride formulation for anesthesia) IV. Digitalis products

* Less than 130 mmHg of mean 24-hour systolic blood pressure and less than 80 mmHg of mean 24-hour diastolic blood pressure at the start of the observation period.
* History of following circulatory-related diseases or symptoms within 24 weeks before start of the observation period.

I. Cardiac disease: Myocardial infarction, coronary artery revascularization II. Cerebrovascular-disease: cerebral infarction, cerebral hemorrhage, transient ischemic attack III. Progressive hypertensive retinopathy: hemorrhage, exudation, or papilledema

* History or complication with the following circulatory-related diseases; Valvular stenosis, atrial fibrillation, pharmacotherapy-required angina, congestion heart failure, or cardiac arrhythmia, or arteriosclerosis obliterans with symptoms of intermittent claudication et al
* Day / night reversal
* History of hypersensitivity or allergy to Azilsartan, Amlodipine, or related drugs
* Participant in any other clinical research
* Pregnant, possible to being pregnant, or lactating woman
* Mal-control of blood pressure during informed consent to taking antihypertensive agent
* Any those the investigator or other researchers consider as unsuitable

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 957 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kazuo Kario, Principal Investigator — Chief Professor of Division of Cardiovascular Medicine, Jichi Medical University
Locations (92):
- Japan (92):
  - Jyuzen General Hospital, Niihama, Aichi-ken
  - Junn Clinic, Tsushima, Aichi-ken
  - Seikei-kai New Tokyo Hospital, Matsudo, Chiba
  - Sanshukai Doi Internal Medicine Clinic, Chikushino-shi, Fukuoka
  - Hakataeki-higashi Clinic, Fukuoka, Fukuoka
  - Ogata Medical Clinic, Fukuoka, Fukuoka
  - Soejima Naika Clinic, Fukuoka, Fukuoka
  - Junshinkai Nakamura Cardiovascular Clinic, Itoshima, Fukuoka
  - Osaki Clinic, Kitakyushu, Fukuoka
  - Osamura Medical Clinic, Kitakyushu, Fukuoka
  - Hoshi General Hospital, Kōriyama, Fukushima
  - Zensyukai Hospital, Maebashi, Gunma
  - Inoue Neurology Clinic, Hiroshima, Hiroshima
  - Oda medical Clinic, Hiroshima, Hiroshima
  - Hakushoukai Sano Hospital, Asahikawa, Hokkaido
  - Jiseikai Higashiasahikawa Hospital, Asahikawa, Hokkaido
  - Koushinkai Shintomi Naika Clinic, Asahikawa, Hokkaido
  - Aoki Clinic, Sapporo, Hokkaido
  - Houwakai Sapporo Hospital, Sapporo, Hokkaido
  - Mitani Clinic, Sapporo, Hokkaido
  - Shinkotoni Family Clinic, Sapporo, Hokkaido
  - Shoureikan Shinsapporo Seiryou Hospital, Sapporo, Hokkaido
  - Tomakomai City Hospital, Tomakomai, Hokkaido
  - Aiseikai PS Clinic, Fukuoka, Hukuoka
  - Hukuyo naika clinic, Itoshima, Hukuoka
  - Asunaro medical Clinic, Kitakyushu, Hukuoka
  - Keiseikai Gohshi Hospital, Amagasaki, Hyōgo
  - Keijukai Itabashi Clinic, Koga, Ibaraki
  - Kamata medical Clinic, Morioka, Iwate
  - Koyokai Hanamure Hospital, Ichikikushikino, Kagoshima-ken
  - Izumi General Medical Center, Izumi, Kagoshima-ken
  - Iroden Clinic, Kamakura, Kanagawa
  - Nagasu Clinic, Kamakura, Kanagawa
  - Himawari-kai Kanagawa Himawari Clinic, Kawasaki, Kanagawa
  - Kawasaki Saiwai Clinic, Kawasaki, Kanagawa
  - Wakoukai Kawasaki Rinko General Hospital, Kawasaki, Kanagawa
  - Hakuai Clinic, Sagamihara, Kanagawa
  - Kaneshiro Diabetes Clinic, Sagamihara, Kanagawa
  - Yamamoto Clinic, Sagamihara, Kanagawa
  - Tsuruma Kaneshiro Diabetes Clinic, Yamato, Kanagawa
  - Furuie Clinic, Yokohama, Kanagawa
  - Minamisawa Clinic, Yokohama, Kanagawa
  - Shintoukai Yokohama Minoru Clinic, Yokohama, Kanagawa
  - Shuyu-kai Kikuchi Clinic, Yokohama, Kanagawa
  - Tani Clinic, Yokohama, Kanagawa
  - Higashikatsuyama Nakazawa Naika Allergy Internal Medicine, Sendai, Miyagi
  - Shinden Higashi Clinic, Sendai, Miyagi
  - Kosei-kai Nijigaoka Hospital, Nagasaki, Nagasaki
  - Meiwakai Izaki Clinic, Ōmura, Nagasaki
  - Shoninkai Shonin Hospital, Beppu, Oita Prefecture
  - Seizenkai Okayama Saidaiji Hospital, Okayama, Okayama-ken
  - Yasuda Clinic, Okayama, Okayama-ken
  - Hirano Doujinkai Tsuyama Daiichi Hospital, Tsuyama, Okayama-ken
  - Taira Hospital, Wake-gun, Okayama-ken
  - AMC Nishiumeda Clinic, Osaka, Osaka
  - Kouseikai Chimori Medical Clinic, Osaka, Osaka
  - Tenjin Tanaka Internal Medicine Clinic, Takatsuki, Osaka
  - Enomoto Clinic, Ageo, Saitama
  - Kazo Minami Clinic, Kazo, Saitama
  - Asukurepiosu Enomoto Clinic, Kumagaya, Saitama
  - Shibuya Clinic, Kumagaya, Saitama
  - H&Y Akimoto Naika Clinic, Saitama, Saitama
  - Shiseidou Tomita Hospital, Saitama, Saitama
  - Takahashi Clinic, Saitama, Saitama
  - Genkikai Wakasa Clinic, Tokorozawa, Saitama
  - JA Shizuoka Kohseiren Enshu Hospital, Hamamatsu, Shizuoka
  - Shimoda Medical Center, Shimoda, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - DIC Utsunomiya Central Clinic, Utsunomiya, Tochigi
  - Nippori Clinic, Arakawa-ku, Tokyo
  - Eireikai Niwa Family Clinic, Chōfu, Tokyo
  - Keiyu Clinic, Chuo-ku, Tokyo
  - Nihonbashikabutocho Nakajima Clinic, Chuo-ku, Tokyo
  - Tokyo Center Clinic, Chuo-ku, Tokyo
  - Taiseikai Seikoudou Clinic, Edogawa-ku, Tokyo
  - Hirookai Kanbara Clinic, Koto-ku, Tokyo
  - Ono Medical Clinic, Koto-ku, Tokyo
  - Sawai Medical Clinic, Koto-ku, Tokyo
  - Shinsei-kai Kameido Ekimae Ckinic, Koto-ku, Tokyo
  - Shinseikai Kameido Minami-guchi Clinic, Koto-ku, Tokyo
  - Kamada Clinic, Mitaka, Tokyo
  - Mitaka Health Care Clinic, Mitaka, Tokyo
  - Murenosato Clinic, Mitaka, Tokyo
  - Shirayurikai Swing Bldg Nozaki Clinic, Musashino, Tokyo
  - Kenkoukan Suzuki Clinic, Ōta-ku, Tokyo
  - Keichikai Shimokitazawa Tomo Clinic, Setagaya-ku, Tokyo
  - Ishinkai Oda Clinic, Shinjuku-ku, Tokyo
  - Ryousyukai Kanauchi Medical Clinic, Shinjuku-ku, Tokyo
  - Shingakai MaO Clinic, Suginami-ku, Tokyo
  - Keiseikai Otsuka Kita-guchi Clinic, Toshima-ku, Tokyo
  - Fujino Clinic, Ube, Yamaguchi
  - Hirokai Higashikatsura Medical Clinic, Tsuru, Yamanashi

REFERENCES:
- [Derived] Kario K, Hoshide S. Age-related difference in the sleep pressure-lowering effect between an angiotensin II receptor blocker and a calcium channel blocker in Asian hypertensives: the ACS1 Study. Hypertension. 2015 Apr;65(4):729-35. doi: 10.1161/HYPERTENSIONAHA.114.04935. Epub 2015 Feb 2. PMID 25646296

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was performed at hospital and clinic
Pre-assignment Details: 957 patients was enrolled in this study. In run-in period, 239 patients were withdrawn.
Period: Overall Study
Arm/Group | Azilsartan | Amlodipine
Started | 359 | 359
Completed | 332 | 336
Not Completed | 27 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azilsartan | Amlodipine | Total
Number analyzed (Participants) | 359 | 359 | 718
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (12) | 61 (12) | 61 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157 | 157 | 314
  Male | 202 | 202 | 404
Region of Enrollment [Number; unit: participants]
  Japan | 359 | 359 | 718
Clinic SBP [Mean (Standard Deviation); unit: mmHg] | 149.6 (10.2) | 150.5 (10.2) | 150.1 (10.2)
Clinic DBP [Mean (Standard Deviation); unit: mmHg] | 90.3 (9.4) | 89.8 (9.6) | 90.1 (9.5)
24-hour SBP [Mean (Standard Deviation); unit: mmHg] | 150.6 (13.0) | 152.4 (13.7) | 151.5 (13.4)
24-hour DBP [Mean (Standard Deviation); unit: mmHg] | 89.3 (8.6) | 90.4 (9.3) | 89.8 (9.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Nocturnal Systolic Blood Pressure Level
Description: Change at the end of a treatment period (Week 8) from the beginning point of an observation period
  *Nocturnal systolic blood pressure level: the mean value of systolic arterial pressure during night (during sleeping)
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan | Amlodipine
Number analyzed (Participants) | 359 | 359
mmHg | -12.6 (15.4) | -17.5 (14.0)

2. Secondary Outcome: Change in the Absolute Value in Difference With Targeted Value* (15 Percent) of Nocturnal Systolic Blood Pressure Fall**
Description: Change from the start of the run-in period (Week -1) at the end of the treatment period (Week 8) *The targeted value has been set as the median of the dipping rate, normal type of nocturnal blood pressure variation, rate of nocturnal blood pressure fall (10-20 percent)
  ** Rate of nocturnal blood pressure fall: calculated as (awake SBP-sleep SBP)/awake SBP
Time Frame: Baseline and 8 weeks
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Azilsartan | Amlodipine
Number analyzed (Participants) | 321 | 331
mmHg
  riser | -7.3 [-10.0 to -4.5] | -10.1 [-13.5 to -6.6]
  non-dipper | -0.7 [-1.9 to 0.6] | -2.1 [-3.1 to -1.1]
  dipper | 4.5 [3.6 to 5.4] | 3.1 [2.3 to 3.8]
  extreme dipper | -1.9 [-3.9 to 0.1] | -3.1 [-4.9 to -1.2]

3. Secondary Outcome: Change in Nocturnal Diastolic Blood Pressure Level
Description: Change from the start of the run-in period (Week -1) at the end of the treatment period (Week 8)
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan | Amlodipine
Number analyzed (Participants) | 359 | 359
mmHg | -7.1 (8.5) | -8.9 (7.9)

4. Secondary Outcome: Change in 24-hour Mean Systolic Blood Pressure Level
Description: Change from the start of the run-in period (Week -1) at the end of the treatment period (Week 8)
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan | Amlodipine
Number analyzed (Participants) | 359 | 359
mmHg | -14.0 (13.3) | -17.5 (11.5)

5. Secondary Outcome: Change in 24-hour Mean Diastolic Blood Pressure Level
Description: Change from the start of the run-in period (Week -1) at the end of the treatment period (Week 8)
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan | Amlodipine
Number analyzed (Participants) | 359 | 359
mmHg | -7.9 (7.5) | -8.9 (6.3)

ADVERSE EVENTS:
Time Frame: 8weeks
Arm/Group | Azilsartan | Amlodipine
Serious Adverse Events (participants affected / at risk) | 0/359 | 5/359
Other Adverse Events (participants affected / at risk) | 91/359 | 77/359
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan (N=359) | Amlodipine (N=359)
Diverticulitis (Gastrointestinal disorders) | 0 | 1
Stroke (Vascular disorders) | 0 | 1
Nettle rash (Skin and subcutaneous tissue disorders) | 0 | 1
Cancer (Gastrointestinal disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan (N=359) | Amlodipine (N=359)
Infectious disease (Infections and infestations) | 30 | 34
Other (Musculoskeletal and connective tissue disorders) | 62 | 49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PIs is that PIs must get approval about publish by study director(Kazuo Kario).